CLINICAL TRIAL: NCT01738841
Title: Post-marketing Surveillance Study of GSK Biologicals' Live, Attenuated Measles, Mumps, Rubella and Varicella Vaccine, Priorix-Tetra, Following a Single Vaccine Dose Given According to Local Prescribing Information in the Philippines
Brief Title: Safety Study of Measles-Mumps-Rubella-Varicella (MMRV) Vaccine, Priorix-Tetra™ in Children Living in the Philippines
Status: Withdrawn | Type: Observational
Why Stopped: Local authorities no longer require routine PMS studies; GSK does not believe the study would add meaningfully to the safety data already available for MMRV.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114229
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Mumps; Rubella; Measles; Varicella
Keywords: Combined measles-mumps-rubella-varicella vaccine; Priorix-Tetra™; MMRV; children; Post-marketing surveillance; Philippines
MeSH Terms: conditions — Mumps; Rubella; Measles; Chickenpox | interventions — Priorix-Tetra vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort Group: Children aged 12 months to 12 years will receive Priorix-Tetra as prescribed by the physician.
  Interventions: Biological: Priorix-Tetra™; Other: Safety data collection

INTERVENTIONS:
Biological: Priorix-Tetra™ — Single dose, subcutaneous injection
Other: Safety data collection — Recording of adverse events, using diary cards

SUMMARY:
This study will collect data on the safety of the MMRV vaccine (Priorix-Tetra™) used in routine practice in children aged 12 months to 12 years living in the Philippines.

DETAILED DESCRIPTION:
The participating physicians will enroll only those subjects for whom they would prescribe Priorix-Tetra in the course of their normal clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Male or female subjects living in the Philippines between, and including, the ages of 12 months and 12 years at the time of the vaccination.
* Female subjects of child bearing potential may be enrolled in the study, if the subject:

  * has agreed to be abstinent or practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 3 months after completion of the vaccination.

Exclusion Criteria:

* Child in care.
* Any contraindications to vaccination as stated in the Prescribing Information.
* Acute, severe febrile illness at the time of enrollment. The presence of a minor infection, such as a cold, will not exclude the subject from the study.
* Previous receipt of a measles, mumps, rubella and/or varicella-virus containing vaccine less than 3 months prior to study entry.
* Previous enrolment in this trial.
* Subjects with impaired immune function, including primary or secondary immunodeficiencies based on medical history.
* History of hypersensitivity to any component of the vaccine.
* History of hypersensitivity following previous administration of measles, mumps, rubella and/or varicella-virus containing vaccines.
* Receipt of human gamma globulins or a blood transfusion within 3 months prior to study entry.
* Hypersensitivity to latex.
* Pregnant or lactating female.

Ages: 12 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 12 months to 12 years living in Philippines will receive Priorix-Tetra as prescribed by the physician.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Grade 3 adverse events (AEs) with a causal relationship to vaccination | Between Day 0 and Day 42

SECONDARY OUTCOMES:
Occurrence of Grade 3 AEs | Between Day 0 and Day 42
Occurrence of medically-attended AEs | Between Day 0 and Day 42
Occurrence of Serious Adverse Events (SAEs) | From the time of vaccination (Week 0) to study end (Week 6)
Occurrence of febrile convulsions | Between Day 0 and Day 42

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline